CLINICAL TRIAL: NCT06217978
Title: The Image Characteristics of Epiploic Appendagitis on Ultrasound and Computed Tomography
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202111032RIND
Record Dates: First submitted 2023-12-24; First posted 2024-01-23 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2023-12

CONDITIONS: Epiploic Appendagitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Epiploic appendagitis is a benign and self-limited condition. However, incorrect diagnosis might lead to unnecessary admission, antibiotics use, or operation.

The patient having epiploic appendagitis usually appeared at our emergency room with the complaint of abdominal pain. There are numerous differential diagnoses when it comes to abdominal pain. Epiploic appendagitis might happen at any part of the colon. Therefore, diverticulitis or appendicitis might be suspected at the first moment. However, epiploic appendagitis might present different image characteristics besides diverticulitis or appendicitis under ultrasound or computed tomography. Some small case number retrospective reviews suggested that epiploic appendagitis was a 2-3cm, oval-shaped, fat density mass with fat stranding under the computed tomography. Under ultrasound, a noncompressible, hyperechoic ovoid mass might impress epiplopic appendagitis.

As ultrasound has become a more and more useful and convenient diagnostic tool in the emergency room, we could diagnose epiploic appendagitis quickly and correctly to reduce unnecessary management.

We would like to compare the image characteristics between the ultrasound image and the computed tomography image to help us to diagnose appendigitis with ultrasound in the future. Furthermore, we would also like to compare the computer tomography image of epiploic appendagitis in different locations.

DETAILED DESCRIPTION:
The incidence of the epiploic appendagitis is unknown. However, some of the patients were first to be suspected to have appendicitis or diverticulitis, the percentages were 2% to 7% and 0.3% to 1 %, respectively. Epiploic appendages are small outpouchings of fat-filled structures presented on the colon's surface. The adult usually has 50-100 appendages along the entire colon. Epiploic appendagitis is defined as an ischemic infarction caused by torsion or spontaneous thrombosis of the central draining vein. Epiploic appendagitis is a benign and self-limited condition. However, incorrect diagnosis might lead to unnecessary admission, antibiotics use, or operation.

The patient having epiploic appendagitis usually appeared at our emergency room with the complaint of abdominal pain. There are numerous differential diagnoses when it comes to abdominal pain. Epiploic appendagitis might happen at any part of the colon. Therefore, diverticulitis or appendicitis might be suspected at the first moment. However, epiploic appendagitis might present different image characteristics other than diverticulitis or appendicitis under ultrasound or computed tomography. Some small case number retrospective reviews suggested that epiploic appendagitis was a 2-3cm, oval-shaped, fat density mass with fat stranding under the computed tomography. Under ultrasound, a noncompressible, hyperechoic ovoid mass might impress epiplopic appendagitis.

As ultrasound has become a more and more useful and convenient diagnostic tool in the emergency room, we could diagnose epiploic appendagitis quickly and correctly to reduce unnecessary management.

We would like to compare the image characteristics between the ultrasound image and the computer tomography image to help us to diagnose appendigitis with ultrasound in the future. Furthermore, we would also like to compare the computed tomography image of epiploic appendagitis in different locations.

ELIGIBILITY:
Inclusion Criteria:

* epiploic appendagitis was diagnosed by ultrasound or CT without other bowel pathology.

Exclusion Criteria:

* Secondary epiploic appendagitis due to appendicitis, diverticulitis or other pathology.

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients admitted to the National Taiwan University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-05-31 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
The location of epiploic appendagitis | 3 weeks
  The location of epiploic appendagitis by ultrasound and CT

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Ching Lien, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Wan-Ching Lien, Taipei, None Selected, Taiwan

IPD SHARING:
Plan to Share IPD: No